CLINICAL TRIAL: NCT01661166
Title: A Phase IV, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study of the Effects of Fesoterodine in Men at High Risk for Overactive Bladder/Detrusor Overactivity Post Robotic-Assisted Laparoscopic Prostatectomy )
Brief Title: A Study of Effects of Fesoterodine in Men at High Risk for Overactive Bladder/Detrusor Overactivity Post Robotic-Assisted Lap. Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPCC 15810
Record Dates: First submitted 2012-07-18; First posted 2012-08-09 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Prostate Adenocarcinoma
Keywords: Male adult subjects; aged 30-90 years; RARP; American Urological Association symptom score greater than 7 will be included
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fesoterodine 4mg (Experimental): Fesoterodine 4mg, Oral once daily for three months
  Interventions: Drug: Fesoterodine
- Placebo (Placebo Comparator): Placebo Oral once daily for three months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Fesoterodine — 4 mg
  Arms: Fesoterodine 4mg
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
The investigators will assess the incidence of Overactive Bladder/Detrusor Overactivity (OAB/DO) post-operatively in patients post robotic assisted radical prostatectomy (RARP) and to investigate whether fesoterodine will alter the incidence of OAB/DO in these patients. Additionally, the correlation between OAB symptoms and urodynamic DO will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 30 to 90 years old with prostate adenocarcinoma who have already made their treatment selection of RARP, and only men with an AUA symptom score greater than 7 will be included. All subjects must be able to read and comprehend fully the informed consent.

Exclusion Criteria:

* Men with prostate neoplasms other than adenocarcinoma
* Subjects receiving other treatments for prostate cancer will be excluded.
* Any subject with a preexisting bladder disease will be excluded.
* Subjects with acute urinary retention and/or deceased gastrointestinal motility.
* Subjects with glaucoma.
* Subjects with hepatic or renal impairment.
* Subjects taking CYP3A4 Inhibitors (e.g.ketoconazole, itraconazole, clarithromycin).
* Subjects with myasthenia gravis
* Subjects who are unwilling or unable to complete the subject questionnaires
* Subjects, who in the opinion of the investigator, would be non-compliant with the majority of the visits scheduled or study procedures.

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States